CLINICAL TRIAL: NCT06916182
Title: Evaluation of Optic Neuritis Using Synthetic Quantitative MRI
Acronym: QUESTION
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2024_11
Record Dates: First submitted 2025-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: MRI sequence — This sequence is a 2D spin-echo sequence for the generation of synthetic maps

SUMMARY:
Inflammatory optic neuropathy (optic neuritis) is an acute condition that can affect the optic nerve along its entire course.

It is a rare event, with a prevalence of up to 5 cases per 100,000 people per year, predominantly affecting young individuals (18-50 years old), primarily Caucasian and female. The causes of optic neuropathy are diverse, with the most common being multiple sclerosis, which is the revealing condition in nearly 30% of cases.

MRI is an integral part of the initial assessment of optic neuritis, in conjunction with clinical examination, laboratory tests, and OCT (optical coherence tomography). It plays a crucial role in the acute management of this condition, particularly by guiding the etiological diagnosis and helping adapt the therapeutic approach accordingly.

The establishment of objective and reliable MRI prognostic markers could allow for more precise immediate therapeutic adjustments, thereby improving the prognosis of this potentially severe and debilitating disease, whose treatment itself is not without risks. Indeed, determining the appropriate corticosteroid dose and deciding whether to combine it with other treatments remains a current clinical challenge.

Despite various publications, MRI prognostic criteria for short- and long-term outcomes of optic neuritis remain unclear. Recent studies using radiomics have shown promising results, but these rely on limited sample sizes. New investigative methods are currently under development in the field of medical imaging, particularly "quantitative MRI."

This approach enables effective analysis through mapping techniques, which generate numerical values compared to predetermined references. For instance:

T1 (or R1) mapping assesses fibrosis and, indirectly, myelination, T2 (or R2) mapping evaluates edema. To our knowledge, this approach has never been studied for the optic nerve.

More recently, the emergence of synthetic imaging has made it possible to generate the previously mentioned R1/R2 maps, along with more conventional weighted images (T1, T2, FLAIR, DP), from a single MRI sequence (2D spin-echo sequence). This sequence provides quantitative values while maintaining a short acquisition time (~5 minutes), which is essential in ophthalmologic imaging, where motion artifacts are frequent.

The goal of this study is to identify prognostic criteria for the evolution of optic neuritis using synthetic quantitative MRI sequences, in the form of threshold numerical values.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with a painful unilateral decrease in visual acuity for less than one month
* Referred for contrast-enhanced MRI imaging
* Explicit consent for participation in the study

Exclusion Criteria:

* Ophthalmological diagnosis other than optic neuritis explaining the symptoms
* Known history of optic neuritis (same eye or contralateral eye)
* Ophthalmological history interfering with the interpretation of ophthalmologic examinations (severe myopia, retinopathy)
* Known glaucoma (same eye or contralateral eye)
* Known diabetes
* Patient under legal protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient requiring an MRI as part of the diagnosis of optic neuritis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
visual function at 4 months (ordinal outcome) | 4 months after inclusion
  Visual function will be categorized into four stages:
  1. Normal visual acuity , normal visual field, and OCT, with no identified sequelae.
  2. Normal visual acuity and visual field, but sequelae identified on OCT (ganglion cells or pRNFL).
  3. Normal visual acuity but an abnormal visual field.
  4. Persistently abnormal visual acuity.
  Definitions:
  Normal visual acuity:
  * For bilateral optic neuritis: visual acuity ≥ 10/10.
  * For unilateral optic neuritis: visual acuity ≥ that of the contralateral (unaffected) eye.
  Normal visual field: Mean deviation (MD) > -3 dB.
  Normal OCT (ganglion cell layer and pRNFL):
  Values within the normal range according to the manufacturer's reference data, adjusted for age.